CLINICAL TRIAL: NCT03485846
Title: Multicenter, Open-label, Phase II Safety and Efficacy Study of All-oral Combination Narlaprevir/Ritonavir and Daclatasvir Administered for 12 Weeks in Patients With Genotype 1b Chronic Hepatitis C
Brief Title: Efficacy and Safety of All-Oral Combination of Narlaprevir/Ritonavir and Daclatasvir in Treatment-Naїve Patients With Chronic Hepatitis C Genotype 1b
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Almedis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJ05013046
Record Dates: First submitted 2018-03-02; First posted 2018-04-02 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Chronic Hepatitis C Genotype 1b
Keywords: hepatitis C; chronic; 1b genotype; oral treatment
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — narlaprevir; Ritonavir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Narlaprevir + Ritonavir + Daclatasvir (Experimental): All of enrolled patients receive equal study therapy with Narlaprevir/Ritonavir/Daclatasvir daily for 12 weeks
  Interventions: Drug: Narlaprevir; Drug: Ritonavir; Drug: Daclatasvir

INTERVENTIONS:
Drug: Narlaprevir — 100 mg, oval shaped, concave, yellow film-coated, tablets taken as 200 mg per os daily
  Other Names: Arlansa
Drug: Ritonavir — 100 mg, tablets, taken as 100 mg per os daily
  Other Names: Norvir
Drug: Daclatasvir — 60 mg, tablets, taken as 60 mg per os daily
  Other Names: Daklinza

SUMMARY:
The purpose of this study is to confirm that combination of Narlaprevir, Ritonavir and Daclatasvir is safe and highly effective regimen in treatment-naїve patients with chronic hepatitis C (HCV) genotype 1b infection.

DETAILED DESCRIPTION:
To evaluate effectiveness and safety of treatment with Narlaprevir, Ritonavir and Daclatasvir combination will be selected 105 treatment-naїve patients with chronic HCV genotype 1b without genetic variants coding for the NS5A-Y93 С/H/N/S and/or L31 F/M/V/I amino acid substitutions, eligible as per protocol criteria.

Each patient will participate in the trial approximately up to 38 weeks:

* 2 weeks are expected for screening
* up to 12 weeks for treatment period
* 24 weeks for follow-up period

During treatment period all patient will receive equal drug combination.

Efficacy and safety parameters will be assessed as per primary and secondary endpoints. Also Ctrough for Narlaprevir and Daclatasvir on day 14 will be evaluated as pharmacokinetic objective.

The results of this study will provide new information about treatment of patients with chronic hepatitis C genotype 1 with Narlaprevir/Ritonavir in combination with Daclatasvir during 12 weeks.

ELIGIBILITY:
Inclusion Criteria -

Subjects who meet all of the following criteria are eligible for participation in the study:

* Are willing and able to provide written informed consent.
* Have confirmed chronic HCV infection as documented by:

  1. positive anti-HCV antibody (Ab) test or
  2. positive HCV RNA or
  3. positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit.
* Have HCV genotype 1b at screening as determined by the Central Laboratory. Any non definitive results must exclude the subject from study participation.
* Minimum HCV-RNA level of ≥10,000 IU at baseline.
* No evidence of cirrhosis; availability at Baseline of at least one of the following tests, negative results:

  1. Liver biopsy within 2 years of screening showing absence of cirrhosis;
  2. Fibroscan with a result of ≤ 12.5 kPa within 6 months of baseline/Day1;
  3. FibroTest score of ≤ 0.48 AND APRI of ≤ 1 performed during screening. In the absence of a definitive diagnosis of the presence or absence of cirrhosis by the above criteria, a liver biopsy was required. Liver biopsy results supersede the results obtained by Fibroscan or FibroTest.
* Have a screening electrocardiogram (ECG) without clinically significant abnormalities (P wave < 0.1 s; PQ interval 0,12-0,2 s; QRS complex 0,06-0,1 s; QT interval 0,35-0,49 s).
* Must have the following laboratory parameters at screening:

  1. alanine aminotransferase (ALT) ≤ 10 x the upper limit of normal (ULN);
  2. aspartate aminotransferase (AST) ≤ 10 x ULN;
  3. Hemoglobin ≥ 12g/dL for male, ≥ 11g/dL for female subjects;
  4. Platelets ≥ 50,000cells/mm3;
  5. International normalized ratio (INR) ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR;
  6. Albumin ≥ 3g/dL;
  7. Direct bilirubin ≤ 1.5 x ULN;
  8. Hemoglobin A1c (HbA1c) ≤ 10%;
  9. Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation;
  10. Have not been treated with any investigational drug or device within 30 days of the screening visit.
* A female subject is eligible to enter the study if it is confirmed that she is:

  1. Not pregnant or nursing;
  2. Of non-childbearing potential (i.e., women who have had a hysterectomy, both ovaries removed, or medically documented ovarian failure, or are postmenopausal women >50 years of age with cessation [for ≥12 months] of previously occurring menses), or
  3. Of childbearing potential (i.e., women who had not had a hysterectomy, both ovaries removed, or medically documented ovarian failure). Women ≤ 50 years of age with amenorrhea are considered to be of childbearing potential. These women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the baseline/Day 1 visit prior to enrollment. They must also agree to one of the following from 3 weeks prior to baseline/Day 1 until 6 months after last dose of the investigational drugs:

     1. Complete abstinence from intercourse. Periodic abstinence from intercourse (e.g., calendar, ovulation, sympto thermal, post-ovulation methods) is not permitted Or
     2. Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from the date of screening until 6 months after the last dose of the investigational drugs:

        * intrauterine device (IUD) with a failure rate of < 1% per year;
        * female barrier method: cervical cap or diaphragm with spermicidal agent;
        * tubal sterilization;
        * vasectomy in male partner; Women of childbearing potential must not rely on hormone-containing contraceptives as a form of birth control during the study. Female subjects using a hormone-containing contraceptive prior to screening must stop their contraceptive regimen use from the date of screening until 6 months after their last dose of investigational drugs.
* All male study participants must agree to consistently and correctly use a condom, while their female partner agrees to use either 1 of the non hormonal methods of birth control listed above or a hormone-containing contraceptive listed below, from the date of screening until 6 months after their last dose of investigational drugs:

  * implants of levonorgestrel;
  * injectable progesterone;
  * oral contraceptives (either combined or progesterone only);
  * contraceptive vaginal ring;
  * transdermal contraceptive patch;
* Male subjects must agree to refrain from sperm donation for at least 6 months after the last dose of investigational drugs.
* Are in generally good health as determined by the investigator.
* Are able to comply with the dosing instructions for study drug administration and are able to complete the study schedule of assessments.

Exclusion Criteria -

Subjects with any of the following are not eligible for participation in the study:

* Had prior exposure to IFN, RBV, or other approved or experimental DAA targeting the HCV.
* Had prior exposure to amiodarone within 24 months before the screening
* Are pregnant or nursing female or male with pregnant female partner.
* Сhronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, α1-antitrypsin deficiency, cholangitis).
* Are infected with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
* Have history of malignancy diagnosed or treated within 5 years; subjects under evaluation for malignancy are not eligible.
* Have chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent > 10 mg/day).
* Have clinically relevant drug or alcohol abuse within 12 months of screening. A positive drug screen must exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the investigator.
* Have excessive alcohol consumption, defined as more than 3 drinks on any single day and more than 7 drinks per week for females, and > than 4 drinks on any single day and more than 14 drinks per week for males.
* Have history of solid organ transplantation.
* Have history of clinically significant illness or any other major medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol by Investigators' opinion.
* Have history of a gastrointestinal disorder (or postoperative condition) that can interfere with the absorption of the study drug.
* Have history of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
* Usage of any prohibited concomitant medications as described in the protocol (list of drugs with expected drug-drug interactions due to concomitant ritonavir usage)
* Have known hypersensitivity to the study investigational medicinal product, the metabolites, or formulation excipients.
* Chronic HCV genotype 1b-infected participant who has the presence of genetic variants coding for the NS5A-Y93 С/H/N/S and/or L31 F/M/V/I amino acid substitutions at Screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieved Sustained Virologic Response (SVR12) | Week 12 of follow-up period
  SVR12 - Undetectable HCV RNA by lower limit of detection (LOD) 12 weeks following the end of treatment

SECONDARY OUTCOMES:
The proportion of patients achieved Sustained Virologic Response (SVR24) | Week 24 of follow-up period
  SVR24 - Undetectable HCV RNA by (LOD) 24 weeks following the end of treatment
The proportion of patients achieved End of Treatment Response (ETR) | Week 12 of treatment
  ETR - HCV RNA < LOD at the treatment end
The proportion of patients achieved Sustained Virologic Response (SVR4) | Week 4 of follow-up period
  SVR4 - HCV RNA < LOD 4 weeks after the end of treatment
The proportion of patients developed Viral Breakthrough | Week 12 of treatment
  Viral Breakthrough - Greater than or equal to 1 log10 increase in HCV-RNA above nadir, or detectable HCV-RNA, while on treatment after an initial drop below detection
The proportion of patients Relapsed | Week 12 of follow-up period
  Relapse - HCV RNA undetectable by LOD at the end of treatment with subsequent detectable HCV RNA at the end of the follow-up period (week 12)

OTHER OUTCOMES:
Number of patients with Adverse Events | From initiation of treatment up to week 24 of follow-up period
Number of patients with Serious Adverse Events | From initiation of treatment up to week 24 of follow-up period
Number of patients with Adverse Event leading to permanent discontinuation of the studying treatment regimen | From initiation of treatment up to week 24 of follow-up period
Number of patients with changes in vital signs | From initiation of treatment up to week 24 of follow-up period
Number of patients with abnormal laboratory values | From initiation of treatment up to week 24 of follow-up period
Pharmacokinetics - Ctrough | Day 14 of treatment
  Pre-dose plasma concentrations of Narlaprevir and Daclatasvir

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (4):
- Russia (4):
  - FBIS CSRI of Epidemiology of Federal Service on Customers, Moscow
  - SBEI HPE Moscow State Medical and Dental University n.a. A.I. Evdokimov of Ministry of Health of Russia, Moscow
  - SBHI of Moscow "City Clinical Hospital #24", Moscow
  - St. Petersburg SBHI Center of Prevention and Fight against AIDS and Infection Diseases, Saint Petersburg